CLINICAL TRIAL: NCT03747601
Title: The Development and Human Translation of Temporal Interference Brain Stimulation
Brief Title: Temporal Interference Brain Stimulation
Acronym: TI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Daniel Press, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018P000603
Record Dates: First submitted 2018-09-19; First posted 2018-11-20 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Temporal Interference (TI) Stimulation (Experimental): Temporal Interference stimulation applied to the head via standard electrodes
  Interventions: Device: Temporal Interference (TI) Stimulation

INTERVENTIONS:
Device: Temporal Interference (TI) Stimulation — 2-4 Temporal Interference stimulation sessions. The device is an experimental non-invasive electrical brain stimulator that functions similar to existing non-significant risk devices for electrical stimulation, including human non-invasive brain stimulation. Briefly, the device produces alternating current electrical stimulation in a kilohertz (kHz) range and results in less net charge applied within the brain. The device is powered by rechargeable 20 volt (V) battery (i.e. there is no connection to building power supply). The current is hardwired and limited to 5 milliamp (mA) via internal resistors. It includes extra safety features such as onboard fuses to limit any abrupt high current, and an emergency stop button which effectively insulates the subject and resets the device. The device was tested and characterized at all the required load conditions.

SUMMARY:
The primary aim of this study is to translate temporal interference (TI) stimulation methodology into humans and examine its safety, feasibility, steerability, and focality. In the proposed early phase human experiment, the ability to apply TI stimulation will be assessed along spatial dimensions to selectively modulate neural activity and assess the feasibility of selective targeting deep brain structures without exciting overlaying cortex. The overall goal of the study is to advance TI methodology and its translation to humans.

The specific aims in this study are to

* Assess the safety of TI stimulation.
* Assess the feasibility, focality, and steerability of TI stimulation by selectively modulating activity in subregions of a cortical area (calcarine cortex)

It is hypothesized that TI stimulation can be used to impact different regions of the visual field that are represented within the calcarine fissure of the human brain.

It is hypothesized that TI will be well tolerated by human subjects and side effects will be consistent with other forms of transcranial electric current stimulation (tES).

DETAILED DESCRIPTION:
This is an investigational early phase testing of temporal interference (TI) stimulation in humans. The overall aim of the study is to assess the safety, feasibility, focality, and steerability of TI stimulation by selectively modulating activity in subregions of a cortical area (calcarine cortex - the primary visual cortex)

Healthy subjects who meet inclusion and exclusion criteria will be entered into the study. The study will recruit up to 20 subjects with the aim to complete 12 subjects.

Study Visits:

The study will consist of up to 6 study visits. The screening and baseline visit, the MRI visit, and up to 4 TI study. The screening and baseline visit and TI visits will occur at Beth Israel Deaconess Medical Center in the Berenson-Allen Center. The MRI visit will take place at the Boston University Cognitive Neuroimaging Center. After Informed Consent is obtained, the following screening and baseline procedures will be completed:

* Inclusion and exclusion criteria review
* Subject demographics
* Handedness assessment
* Medical history and medication review
* Physical and Neurological exam conducted by a Neurologist or Neurologic Nurse Practitioner
* Baseline perimetry assessment
* Baseline EEG
* The Mini International Neuropsychiatric Interview (MINI) assessment
* All female subjects will undergo a pregnancy test and pregnant women will be excluded
* Screening for retinotopic mapping - assessing the participant's ability to hold fixation with their eyes for experimental trials
* MRI safety review

The MRI session will take place at the Boston University Cognitive Neuroimaging Center under a Boston University submitted and approved protocol that is specific to this study. An MRI scan of the brain will be conducted while the participant views visual stimuli to obtain each individual's retinotopic map. This data will be provided to the study team at Beth Israel Deaconess Medical Center (BIDMC) to conduct the study visit and for analysis.

Each subject will then undergo up to 4 TI stimulation sessions (2 minimum) separated by at least 2 days to minimize the risk of carry over effects of the stimulation. In each visit, the participant will receive TI stimulation to one of four regions of retinotopic representation in the calcarine fissure:

1. peripheral visual field in the deep region of the fissure
2. foveal visual field in the polar region of the fissure
3. superior quadrant of the visual field in the lower bank of the fissure
4. inferior quadrant of the visual field in the upper bank of the fissure The cortical targets will be defined by electrical field modelling that will be used to optimize the electrode placement. Regions #1 and #2 will be stimulated in the first two visits with the order of stimulation regions to be counterbalanced between participants. If an effect is noted, participants will be asked to complete the additional 2 visits in which regions #3 and #4 will be stimulated.

Each visit will consist of up to 4 blocks of stimulation paired with a visual discrimination task and assessment of visual disturbance with an Amsler grid. The stimulation blocks will each be completed at a different frequency - a control stimulation where TI visual effect is not anticipated (e.g 2 or 20 hertz (Hz)), a no offset stimulation (e.g. matched carrier stimulation frequencies such as no envelope modulation is anticipated) and up to 2 frequencies ranging from 8 to 12. The most common signal from visual cortex during wakeful relaxation is in the frequency range (8-12 Hz). It is hypothesized that TI with a residual effective stimulation frequency of 1-20 Hz will be ideally suited for activation of the targeted visual cortex.

Participants will be monitored throughout he visit for any adverse effects and a tES side-effect questionnaire will be administered at the beginning and end of each stimulation visit to additionally track any adverse effects. Although any visual disruption induced by the stimulation is expected and anticipated to be transient in nature, a visual perimetry assessment will be completed to compare to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* 18-35 years of age
* Normal vision
* Right handed

Exclusion Criteria:

* Corrected-to-Normal vision, or visual impairment.
* Any current or past history of a psychiatric disorder
* Any current or past history of neurological disorders or acquired neurological disease (e.g. stroke, traumatic brain injury), including intracranial lesions
* History of head trauma resulting in prolonged loss of consciousness; or a history of >3 grade I concussions
* Current history of poorly controlled headaches including intractable or poorly controlled migraines
* Any systemic illness or unstable medical condition that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG, or family history of treatment resistant epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Possible pregnancy. All female participants of child bearing age are required to have a pregnancy test
* Any metal in the brain, skull or elsewhere unless approved by the responsible MD
* Any medical devices (i.e. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagal nerve stimulator) unless otherwise approved by the responsible MD
* Substance abuse or dependence within the past six months
* Pregnancy; all female participants of child bearing age will be required to have a pregnancy test; any participant who is pregnant will not be enrolled in the study.
* Not on any medications with the exception of birth control unless approved by the responsible MD.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 enrolled participants did not receive the intervention due to early termination of the study due to COVID.
Period: Overall Study
Arm/Group | Temporal Interference (TI) Stimulation
Started | 8
Completed | 4
Not Completed | 4
Not completed — COVID halt to visits | 4

BASELINE CHARACTERISTICS:
Population: number of participants enrolled in the study
Groups:
- Temporal Interference (TI) Stimulation: Temporal Interference stimulation applied to the head via standard electrodes
  Temporal Interference (TI) Stimulation: 1-4 Temporal Interference stimulation sessions. The device is an experimental non-invasive electrical brain stimulator that functions similar to existing non-significant risk devices for electrical stimulation, including human non-invasive brain stimulation. Briefly, the device produces alternating current electrical stimulation in a kilohertz (kHz) range and results in less net charge applied within the brain. The device is powered by rechargeable 20 volt (V) battery (i.e. there is no connection to building power supply). The current is hardwired and limited to 5 milliamp (mA) via internal resistors. It includes extra safety features such as onboard fuses to limit any abrupt high current, and an emergency stop button which effectively insulates the subject and resets the device. The device was tested and characterized at all the required load conditions.
Arm/Group | Temporal Interference (TI) Stimulation
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Change in Their Visual Field
Description: Number of participants who had a change in their visual field (scitoma) as assessed by a neurophthalmologist.
Time Frame: Immediately after intervention
Population: Other 4 were not able to complete visits due to Covid
Measure: Count of Participants; unit: Participants
Arm/Group | Temporal Interference (TI) Stimulation
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Temporal Interference (TI) Stimulation
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03747601/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT03747601/ICF_001.pdf